CLINICAL TRIAL: NCT06949995
Title: Effects of Blood Flow Restriction on Post-Exercise Recovery in Amateur Runners: A Stratified Randomized Controlled Trial
Brief Title: Effects of Blood Flow Restriction on Post-Exercise Recovery in Amateur Runners
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, Principal investigator, Paulista University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 84324824.9.0000.5402
Record Dates: First submitted 2025-04-09; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Recovery Methods; Recovery Time
Keywords: Running; physiological stress; functional physical performance; post-exercise recovery techniques; blood flow restriction therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active Recovery and Blood Flow Restriction (Experimental): Participants will undergo baseline assessments, followed by a muscle stress protocol. After that, they will perform 10 minutes of active recovery (AR) using a blood flow restriction cuff at 60% of total occlusion pressure
  Interventions: Device: Active Recovery with Blood Flow Restriction
- Active Recovery (Active Comparator): Participants will undergo baseline assessments, followed by a muscle stress protocol. After that, they will perform 10 minutes of active recovery (AR) without any restriction.
  Interventions: Other: Active Recovery
- Control (No Intervention): Participants will undergo baseline assessments, followed by a muscle stress protocol. After that, they will undergo 10 minutes of absolute rest, without any movement or intervention.

INTERVENTIONS:
Device: Active Recovery with Blood Flow Restriction — 10-minute active recovery protocol performed with blood flow restriction using a pneumatic cuff set at 60% of the participant's total occlusion pressure.
  Arms: Active Recovery and Blood Flow Restriction
Other: Active Recovery — 10-minute active recovery protocol.
  Arms: Active Recovery

SUMMARY:
Street running has become an increasingly popular sport. As a result, effective recovery strategies after exercise are essential. In this context, two techniques stand out: one already validated, active recovery (AR), and another with potential, blood flow restriction (BFR). This study aims to investigate whether using both techniques simultaneously can benefit practitioners and improve outcomes compared to complete rest.

DETAILED DESCRIPTION:
This randomized clinical trial aims to evaluate the effects of combining active recovery (AR) and blood flow restriction (BFR) on post-exercise recovery in amateur runners. Thirty-four healthy male participants aged 18-40 years, who run at a pace faster than 5:30 min/km, will be stratified based on their performance in the 3-minute all-out running test and randomly assigned to one of three groups: AR with BFR, AR alone, or passive rest (control). All participants will undergo baseline assessments, followed by a muscle stress protocol, the assigned recovery strategy, and follow-up evaluations immediately, and at 24, 48, 72, and 96 hours post-exercise.

Outcomes include heart rate variability (via RR intervals), muscle soreness (Numeric Rating Scale), recovery perception and discomfort (Likert scale), effort (Borg CR-10), cellular integrity (bioelectrical impedance), pain threshold (pressure algometer), muscle tone, stiffness, and elasticity (myotonometry), muscle power (Squat Jump test), plantar flexor strength (digital dynamometer), and maximal aerobic capacity (3-minute test). Data will be analyzed using descriptive statistics and repeated measures ANOVA, with significance set at p<0.05.

Participants will be duly informed about the procedures and objectives of this study, and after agreeing, they will sign an informed consent form, effectively becoming part of it. In the consent form, participants will be asked if they agree to the use of their data if they choose to withdraw from the study. Participants will also be asked for permission for the research team to share relevant data with people at universities participating in the research or regulatory authorities, where relevant. The study will be sent for consideration and approval to the Research Ethics Committee of FCT/UNESP, Presidente Prudente, SP, Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who present one or more of the following characteristics will not be included:
* 1 presence of any health condition that contraindicates or prevents exercise;
* 2 diabetes and diagnosed high blood pressure;
* 3 inflammatory, psychiatric, cardiovascular and/or respiratory rheumatological disease; - -4 being dependent on alcohol, consuming drugs and/or being a smoker;
* 5 history of knee surgery (e.g., meniscal repair and ligament reconstruction) or recent lower limb musculoskeletal injury that may impair performance during tests or interventions (e.g., muscle injury, tendinopathy, patellofemoral pain and/or back pain column in the last six months);
* 6 use of ergogenic supplements to improve physical performance and/or muscle mass and/or vasoactive medications;
* 7 having one or more risk factors predisposing to thromboembolism

Exclusion Criteria:

* Participants will be excluded from the study if they:
* 1 have a health problem that does not allow them to continue;
* 2 wish to leave the study;
* 3 not sign the consent form

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only individuals assigned male at birth will be included, due to physiological characteristics relevant to the study objectives.
Enrollment: 34 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Isometric strength of the triceps surae | Change from baseline at 96 hours after exercise
  The isometric peak torque of the triceps surae will be measured using a digital handheld dynamometer (DD-300, Instrutherm). Participants will lie in a prone position with the knee flexed at 90°, foot dorsiflexed, and will be instructed to push maximally against the dynamometer. Three attempts will be performed with a 1-minute rest interval. The highest value will be used for analysis.
Aerobic capacity | Change from baseline at 96 hours after exercise
  Aerobic capacity will be evaluated using a 3-minute all-out running test (TM3) on a non-motorized treadmill. After a 5-minute warm-up at 7 km/h, participants will run at maximal effort for 3 minutes. Power and velocity outputs will be recorded by the treadmill's sensors and used to calculate critical power (CP) and critical velocity (CV).
Lower limb muscle power | Change from baseline at 96 hours after exercise
  Muscle power will be assessed through the Squat Jump test using a contact platform (Multisprint). Participants will begin in a 90° knee flexion position (verified with a goniometer), with hands on hips, and will perform a vertical jump without countermovement. Variables to be analyzed will include jump height, modified reactive strength index, jump power, and take-off moment.
Muscle soreness and pain threshold | Change from baseline at 96 hours after exercise
  Muscle soreness will be assessed using a Numeric Pain Rating Scale (0-10). Pain threshold will be measured with a pressure algometer (FPX 50/220; Wagner) at four sites: biceps femoris, rectus femoris, tibialis anterior, and gastrocnemius. Measurements will be recorded in kgf and will not exceed 2.55 kgf.
Perceived exertion, recovery, and discomfort | Change from baseline at 96 hours after exercise
  Perceived exertion, recovery, and discomfort will be measured using the Borg CR-10 scale (0-10). Participants will rate: (1) exertion as whole-body effort, (2) discomfort as muscular sensations in the lower limbs, and (3) recovery as general physical and psychological recovery. Values will be individually recorded at each time point.
Myotonometry | Change from baseline at 96 hours after exercise
  Muscle tone, stiffness, and elasticity will be measured using the MyotonPRO device. The probe will be positioned perpendicularly over the following sites: biceps femoris, rectus femoris, tibialis anterior, and gastrocnemius. The device will apply a 0.18 N pre-load and a 0.40 N impulse to induce tissue oscillation for measurement.
Bioelectrical impedance analysis | Change from baseline at 96 hours after exercise
  Bioimpedance will be measured using a tetrapolar device (BIA Analyzer, 50 kHz, 800 µA). Electrodes will be positioned on the biceps femoris, rectus femoris, tibialis anterior, and gastrocnemius. Analyzed variables will include resistance (R), reactance (Xc), phase angle (PhA), and tolerance ellipse, via Bioscan software.
Heart rate variability (HRV) | Change from baseline at 96 hours after exercise
  HRV will be assessed using a validated monitor (Polar V800). RR intervals will be collected at rest (10 minutes), during a 10-km run, and post-intervention (60 minutes). On other days, collections will last 20 minutes. Participants will be instructed to avoid stimulants during data collection.

OTHER OUTCOMES:
Occlusion pressures (AOP) | Baseline
  To determine the AOP, the Doppler equipment transducer will be used, which will be positioned over the posterior tibial artery to capture the auscultatory pulse. A blood pressure cuff will be fixed to the participant's thigh close to the region of the inguinal fold of the dominant limb, and then with the inflatable region of the cuff on the medial portion of the thigh covering the femoral artery, it will be progressively inflated, waiting 15 seconds every 30 mmHg until the point at which the auscultatory pulse of the tibial artery is interrupted.

CONTACTS AND LOCATIONS:
Locations (1):
- Franciele Marques Vanderlei, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No